CLINICAL TRIAL: NCT02292836
Title: Rosacea Prevalence in General Population - Pilot Study
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: RD.03.SPR.29105
Record Dates: First submitted 2014-10-14; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- rosacea patients: Questionnaire testing on routine dermatologist patient population
  Interventions: Other: Questionnaire testing
- non-rosacea patients: Questionnaire testing on routine dermatologist patient population
  Interventions: Other: Questionnaire testing

INTERVENTIONS:
Other: Questionnaire testing — Questionnaire testing on rosacea and non-rosacea dermatology outpatients

SUMMARY:
The purpose of this study is to test and refine, a subject questionnaire aimed to be used in a general population rosacea prevalence study.

DETAILED DESCRIPTION:
The study will test the subject questionnaire aimed to be used in a full general population prevalence study to screen potential subjects with rosacea.

Questionnaire will be self-administrated to Dermatology outpatients.

Testing will be performed at the practice of 2 Dermatologists experts in rosacea who will evaluate subjects' answers and propose fine-tuning of the questionnaire content, if needed.

ELIGIBILITY:
* Male or Female aged between 18 (or locally accepted majority) and 65 years old both included.
* Subject visiting one of the study dermatology practices for daily care/routine dermatology consultation.
* Subject have to read and sign the approved Informed Consent form prior to any participation in the study,
* Subject willing and capable of cooperating to the extend and degree required by the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rosacea and non-rosacea patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of questions | Day 1
  sensitivity and specificity of each questionnaire key items by comparing subject answers and investigator assessments, as follows: Sensitivity= True Positive/(True Positive+False Negative)
  Specificity= True Negative/ (False Positive+True Negative)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien AUDIBERT, Bsc, Study Director — Galderma R&D
Locations (2):
- Jerry TAN, Windsor, Ontario, Canada
- Mats BERG, Eskilstuna, Sweden